CLINICAL TRIAL: NCT05691803
Title: Understanding Motivation Towards Exercise to Enhance Physical Activity on Prescription Adherence - Feasibility Study
Acronym: UMEPA-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Andreas Hult, Associate Professor, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMEPA01
Record Dates: First submitted 2022-12-21; First posted 2023-01-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity
Keywords: Physical inactivity; Exercise Referral Scheme; Physical activity on Prescription; Exercise intervention; Feasibility study
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A one arm intervention study with allocation to usual care (Physical activty on Prescription) + an exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise intervention (Experimental): Participants are prescribed a Physical activity on Prescription (PaP) which means that they will have a motivational interview with a physiotherapist regarding increased physical activity. The physiotherapist will then prescribe a individualized PaP with the goal to increase weekly physical activity that the participant are instructed to adhere to for the remainder of the study. A follow-up session is also included after 12 weeks.
  Participants are invited to a 12 week exercise intervention at a private fitness center after they have received their PaP. The exercise, including a variety of aerobic and resistance training, is performed in a group setting starting with one session per week for the first three weeks and then two sessions per week for week 4-12. A follow-up session is also included after 12 weeks.
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — The 6 month intervention consists of usual care (PaP) plus an initial 12 weeks of instructor led exercise (described below) followed by a 12 week period in where the participant will have to conduct their physical activity on their own.
  Exercise intervention:
  Participants are invited to a 12 week exercise intervention at a private fitness center after they have received their PaP. The exercise, including a variety of aerobic and resistance training, is performed in a group setting starting with one session per week for the first three weeks and then two sessions per week for week 4-12. A follow-up session is also included after 12 weeks in where a physiotherapist contact the participant and discuss how they will adhere to their Physical activity on prescription.

SUMMARY:
The goal of this clinical trial is to explore feasibility and evaluate methods to investigate changes in physical activity, function and psychometrics in relation to an exercise intervention in physically inactive middle-aged men and women. The main questions it aims to answer are:

* Is the exercise intervention feasible regarding retention and user experience?
* Is the evaluation methods on physical activity, function and psychometrics suitable for the present study?
* Is there an intervention effect in physical activity, function and psychometrics at three and six month post baseline?
* Can barriers and facilitators towards increased physical activity be identified in the two groups of the study?

All participants will first receive standard care for physically inactive patients, i.e. Physical activity on Prescription (PaP), followed by allocation to an exercise intervention (EI) group. The EI group will be offered an additional exercise intervention for 12 weeks consisting of 1-2 training sessions per week of a combination of aerobic and resistance training at a private fitness center.

Feasibility of the exercise intervention will be evaluated based on retention rates and user experience.

Additionally, researchers will assess physical activity, function and psychometrics in the EI group at three and six months to evaluate the suitability of the chosen methods and to get preliminary data on the intervention effect. Finally, interviews with the participants in the control and EI groups will be performed at the end of the study in order to explore barriers and facilitators towards increased physical activity in formally inactive patients.

Edit after registration of the study: Due to a lower number of recruited participants than expected (20 instead of the anticipated 30), the protocol was updated by removing the control group that would initially consist of 10 participants. The remaining 20 participants were all allocated to the exercise intervention group to assess feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive persons as defined as not meeting the current recommendations of at least 150 minutes of moderate to vigorous physical activity per week. This criterion is self-assessed by potential participants.
* Age 40-60 years

Exclusion Criteria:

* Physical disability that affects the ability to perform the exercise intervention.
* Heart failure or severe degenerative disease, e.g. malignant cancer, multiple sclerosis etc.
* Myocardial infarction or stroke during the last 12 months.
* Heart conditions including angina pectoris that is worsened with exercise.
* Neuromuscular, musculoskeletal, or rheumatic conditions that is worsened with exercise.
* Hypertension grade III, i.e. systolic blood pressure above 180 mmHg and/or diastolic blood pressure over 110 mmHg.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Adherence to the exercise intervention | Documented continuously during the 12 week intervention period
  Number of completed training sessions in the exercise intervention group
Retention rate | 3 months post baseline
  The proportion of participants starting the intervention that completes outcome assessment in either group

SECONDARY OUTCOMES:
Time spent in moderate and vigorous physical activity | Baseline, 3 months and 6 months
  Objectively measured physical activity, measured with an accelerometer for 7 consecutive days. Raw data are then recalculated to minutes spent in different intensity zones and finally minutes in moderate and vigorous physical activity are calculated.
Daily step-count | Baseline, 3 months and 6 months
  Objectively measured physical activity, measured with an accelerometer for 7 consecutive days is used to collect step-count which is presented as steps taken per day.
Cardio-respiratory capacity | Baseline, 3 months and 6 months
  Ekblom-Bak cycle ergometer test will be used to assess cardio-respiratory fitness.
Upper limb strength | Baseline, 3 months and 6 months
  Hand grip strength om the non dominant hand is measured with a hand dynamometer to the nearest kg. Three consecutive trials is performed in a seated position with the elbow held at a 90 degree angle and the highest value is recorded. A higher value indicate higher upper limb strength.
Lower limb muscle strength | Baseline, 3 months and 6 months
  Five repetition sit to stand test. From a seated position, the participant is instructed to stand up and then sit down again for a total of five times. The total time of five repetition sit to stand cycles is then recorded in seconds with a stopwatch. A lower total time indicate higher lower limb muscle strength.
Health related quality of life | Baseline, 3 months and 6 months
  RAND-36 health survey will be used (RAND is not an acronym but the name of a research corporation). The RAND-36 survey contains 36 questions belonging to eight health concepts that can be further categorized into two summary scores; physical and mental health. The answers from the survey is re-coded into points in where higher points indicate better perceived health. The points, ranging from 0 to 100, are then presented for the different concepts, the two summary scores and the overall score for the 36 questions.
Self-reported exercise and physical activity | Baseline, 3 months and 6 months
  One question regarding exercise and one question regarding every day physical activity in a typical week. The question regarding exercise comprises 6 answer alternatives ranging from 0 min to more than 120 min per week. The question regarding every day physical activity comprises 7 answer alternatives raging from 0 min to more than 300 min per week. The questions are produced by the Swedish National Board of Health and Welfare.
Motivational stages of self-determination for exercise | Baseline, 3 months and 6 months
  Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) will be used. The questionnaire contains 19 questions, belonging to one of the five categories Amotivation, External regulation, Introjected regulation, Identified regulation and Intrinsic regulation. The scale assesses where a person is on the continuum of self-determination in where higher, positive scores indicate greater relative autonomy; lower, negative scores indicate more controlled regulation.
Confidence in one's own ability to exercise | Baseline, 3 months and 6 months
  The Swedish Exercise Self-Efficacy Scale (ESES-S) will be used. The questionnaire comprises 10 questions on exercise self-efficacy, each with four answer alternatives. The composite score ranges from 10 to 40 and a higher score indicate a higher precised self-efficacy towards exercise.
Basic psychological needs connected to physical activity satisfaction | 3 months and 6 months
  The Basic Psychological Needs in Exercise Scale (BPNES) will be used. This questionnaire contains 12 questions related to one of three basic psychological needs; Autonomy, Competence and Relatedness in the exercise domain. Answers are given on a five point Likert scale and results are presented for the individual needs and as a collective, global need. The maximal score for each question is 5 and the minimal score is 1. Mean values for each need is presented together with a mean score of all 12 questions. A higher score indicate a higher need fulfillment.

OTHER OUTCOMES:
Feasibility of the exercise intervention | 3 months
  Semi-structured qualitative individual interviews will be conducted with the exercise intervention group to explore the user experience of the participants
Exploring barriers and facilitators towards physical activity | 6 months
  Semi-structured qualitative individual interviews will be conducted in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No
Sharing of individual data is not in accordance with the ethical permission granted from the Swedish ethics review authority.